CLINICAL TRIAL: NCT01146678
Title: A Randomized, Cross-over, Open, Euglycemic Clamp Study on the Relative Bioavailability and Activity of 0.6 U/kg Insulin Glargine and 20 μg Lixisenatide, Given as On-site Mix Compared to Separate Simultaneous Injections in Subjects With Type 1 Diabetes Mellitus
Brief Title: Relative Bioavailability and Activity of Different Formulations of Insulin Glargine and Lixisenatide in Patients With Diabetes Mellitus Type 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BDR11578; 2010-019228-30 (EudraCT Number); U1111-1116-8960 (Other: UTN)
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — lixisenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lantus(insulin glargine)/lixisenatide on-site mix (Experimental): Single dose injection of an on site mix of Lantus U100 and lixisenatide (800µg/mL in Lantus U100) at one peri-umbilical site under fasting conditions
  Interventions: Drug: Insulin glargine HOE901; Drug: Lixisenatide AVE0010
- lixisenatide + Lantus (insulin glargine) (Active Comparator): Single dose, separate injection simultaneous injections of Lantus U100 and lixisenatide (100µg/mL) at opposite peri-umbilical sites within 1 minute under fasting conditions
  Interventions: Drug: Insulin glargine HOE901; Drug: Lixisenatide AVE0010

INTERVENTIONS:
Drug: Insulin glargine HOE901 — Pharmaceutical form:solution for injection
  Route of administration: subcutaneous
Drug: Lixisenatide AVE0010 — Pharmaceutical form:solution for injection
  Route of administration: subcutaneous

SUMMARY:
Primary Objective:

* to assess the relative bioavailability of a single dose of insulin glargine (Lantus) and lixisenatide given subcutaneously as on-site mix versus separate and simultaneous injections of each drug

Secondary Objectives:

* to compare the activity of a single dose of insulin glargine and lixisenatide given subcutaneously as on-site mix versus separate and simultaneous injections of each drug
* to assess the safety and tolerability of insulin glargine and lixisenatide given subcutaneously as on-site mix

DETAILED DESCRIPTION:
The study period for one patient is one month in average and it can last up to 7 months (+ 2 weeks) with post-study and follow-up visits

ELIGIBILITY:
Inclusion criteria:

* Subjects with type 1 diabetes mellitus for more than one year with total insulin dose of <1.2 U.kg/day, but otherwise healthy with glycohemoglobin (HbA1c) ≤ 9.0%, stable insulin regimen for at least 2 months prior to study, normal finding in medical history and physical examination.

Exclusion criteria:

* any history or presence of clinically relevant cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic (apart from diabetes mellitus type I), hematological, neurological, psychiatric, systemic (affecting the body as a whole), ocular, gynecologic (if female), or infectious disease; any acute infectious disease or signs of acute illness
* More than one episode of severe hypoglycemia with seizure, coma or requiring assistance of another person during the past 6 months
* Frequent severe headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month)
* Symptomatic hypotension, or asymptomatic postural hypotension defined by a decrease in systolic blood pressure (SBP) equal to or greater than 20 mmHg within three minutes when changing from the supine to the standing position
* Presence or history of a drug allergy to clinically significant allergic disease
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol
* Pregnant or breast feeding women
* Any medication within 14 days before inclusion, or within 5 times the elimination half-life of that drug, whichever the longest and regular use of any medication other than insulins in the last month before study start with the exception of thyroid hormones, lipid-lowering and antihypertensive drugs, and, if female, with the exception of hormonal contraception or menopausal hormone replacement therapy, any vaccination within the last 28 days.
* Positive reaction to any of the following tests: hepatitis B surface (HBs Ag) antigen, antihepatitis B core antibodies (anti-HBc Ab) if compound having possible immune activities, anti-hepatitis C virus (anti-HCV2) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab)
* History of unexplained pancreatitis, chronic pancreatitis and/or pancreatectomy

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Area under the plasma lixisenatide concentration curve (LIX-AUClast) | 1 day (D1 to D2) in the first treatment period and 1 day (D1 to D2) during the second treatment period
Lixisenatide maximum plasma/serum peak concentration (LIX-Cmax) | 1 day (D1 to D2) in the first treatment period and 1 day (D1 to D2) during the second treatment period

SECONDARY OUTCOMES:
Area under the plasma lixisenatide concentration curve (AUC) | 1 day (D1 to D2) in the first treatment period and 1 day (D1 to D2) during the second treatment period
Time to Cmax (Tmax ) for lixisenatide | 1 day (D1 to D2) in the first treatment period and 1 day (D1 to D2) during the second treatment period
Area under the body weight standardized glucose infusion rate curve (GIR) within 24 h (GIR-AUC0-24) | 1 day (D1 to D2) in the first treatment period and 1 day (D1 to D2) during the second treatment period
Time to 50% of the GIR-AUC within 24 h (T50%-GIR AUC0-24) | 1 day (D1 to D2) in the first treatment period and 1 day (D1 to D2) during the second treatment period
Maximum smoothed body weight standardized glucose infusion rate GIRmax | 1 day (D1 to D2) in the first treatment period and 1 day (D1 to D2) during the second treatment period
Time to GIRmax (GIR-Tmax) | 1 day (D1 to D2) in the first treatment period and 1 day (D1 to D2) during the second treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Berlin, Germany